CLINICAL TRIAL: NCT05744622
Title: Clinical Evaluation of Chemically Cured Conventional Glass Ionomer After Light Emitting Diode Radiant Heat Enhancement: A Randomized Controlled Clinical Trial
Brief Title: Clinical Evaluation of Chemically Cured Conventional Glass Ionomer After Light Emitting Diode Radiant Heat Enhancement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Principal Investigator, eman awad, Assistant lecturer operative dentistry department, Suez Canal University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 431/2021
Record Dates: First submitted 2023-02-15; First posted 2023-02-27 (Actual); Last update posted 2023-02-27 (Actual); Status verified 2023-02

CONDITIONS: High Caries Risk Patients

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- chemically cured conventional glass ionomer restorative (Ketac Universal Aplicap) (Experimental): For restoration of M1 group, capsule activation will be performed through loading of the KetacTM Universal AplicapTM GIC capsule into its activator keeping the applicator nozzle closed, using the ball of my hand to depress the activator lever firmly as far as it will go and hold it down for 2 to 4 seconds. Then the capsule will be mixed in a high frequency mixing device for 8 seconds. The mixed capsule will be immediately removed from the mixer and loaded into the AplicapTM Applier then application nozzle will be opened to extrude the mixture directly into the preparation as a single bulk within 1:40 minute. The preliminary contour will be done using a ball burnisher.
  Interventions: Other: KetacTM Universal AplicapTM
- Ketac Universal Aplicap enhanced with light-emitting diode radiant heat (Experimental): Restoration of M2 group will be performed following the same steps which will be carried out for M1 group but the achieved restorations will be enhanced by light-emitting diode radiant heat for 60 seconds
  Interventions: Other: KetacTM Universal AplicapTM with light cure

INTERVENTIONS:
Other: KetacTM Universal AplicapTM — chemically cured conventional GICs
  Arms: chemically cured conventional glass ionomer restorative (Ketac Universal Aplicap)
Other: KetacTM Universal AplicapTM with light cure — chemically cured conventional GICs with light curing enhancement
  Arms: Ketac Universal Aplicap enhanced with light-emitting diode radiant heat

SUMMARY:
Introduction:

Glass ionomer cements (GICs) are widely used in clinical dentistry due to their advantageous properties. However, they present inferior physical and mechanical properties compared to resin composites.

Aim:

Clinical evaluation of chemically cured conventional glass ionomer after light-emitting diode radiant heat enhancement. .

Methodology:

Eighteen healthy patients with 36-second molar teeth will be selected where each patient should have two oclusso- mesial cavities. Standardized oclusso- mesial cavities will be prepared for all the selected teeth, for each patient the first tooth will be restored with chemically cured conventional GICs without any enhancement (M1 group). Meanwhile, the second tooth will be restored by chemically cured conventional GICs that enhanced with radiant heat (LED) (M2 group). functional and biological criteria of each restoration will be clinically evaluated at 4 time points

DETAILED DESCRIPTION:
Introduction:

Glass ionomer cements (GICs) are widely used in clinical dentistry due to their advantageous properties. However, they present inferior physical and mechanical properties compared to resin composites. Various techniques have been suggested to improve properties of conventional GICs such as radiant heat transfer by Light Emitting Diode (LED) or lasers, ultrasonic energy transfer also using of (CaCl2) solution.

Aim:

Clinical evaluation of chemically cured conventional glass ionomer after light-emitting diode radiant heat enhancement. .

Methodology:

Eighteen healthy patients with 36-second molar teeth will be selected where each patient should have two oclusso- mesial cavities. Standardized oclusso- mesial cavities will be prepared for all the selected teeth, for each patient the first tooth will be restored with chemically cured conventional GICs without any enhancement (M1 group). Meanwhile, the second tooth will be restored by chemically cured conventional GICs that enhanced with radiant heat (LED) (M2 group). functional and biological criteria of each restoration will be clinically evaluated immediately after restoration (T0), six months later (T1), and after 12 months (T2) using Federation Dentaire International (FDI) criteria for assessment of dental restorations.

ELIGIBILITY:
Inclusion Criteria:

1. Age group 21 - 45 years.
2. Both males and females will be included.
3. Ability to return for periodic follow-up (good general health).
4. Only co-operative patients.
5. Vital upper or lower carious posterior teeth.

Exclusion Criteria:

1. Teeth with any pathologic pulpal disease.
2. Teeth with previous restorations
3. Teeth with surface loss due to attrition, erosion, abrasion, or abfraction.
4. Patients with severe or chronic periodontitis.
5. Patients have allergy to the materials used in this trial. 6- Nonfunctioning teeth with no opposing dentition.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2021-02-20 (Actual); Primary Completion 2022-02-20 (Actual); Study Completion 2022-05-22 (Actual)

PRIMARY OUTCOMES:
Clinical performance of biological properties | 12 months
  Clinical performance of biological properties according to FDI criteria
Clinical performance of Functional properties | 12 months
  Clinical performance of Functional properties according to FDI criteria

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of dentistry, Suez Canal university, Ismailia, Egypt

IPD SHARING:
Plan to Share IPD: No